CLINICAL TRIAL: NCT01716754
Title: A Multi-center, Randomized, Double-blind, Placebo and Active-controlled Study With Exploratory Dose-ranging to Investigate the Efficacy and Safety of 16 Weeks Treatment With Subcutaneous (s.c.) QGE031 in Asthma Patients Not Adequately Controlled With High-dose Inhaled Corticosteroids and Long Acting β2-agonists
Brief Title: Efficacy and Safety of QGE031versus Placebo and Omalizumab in Patients Aged 18-75 Years With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQGE031B2201; 2012-002298-69 (EudraCT Number)
Record Dates: First submitted 2012-10-19; First posted 2012-10-30 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: asthma; asthma control; allergy; atopic; IgE; double-blind; placebo; omalizumab
MeSH Terms: conditions — Asthma; Hypersensitivity | interventions — ligelizumab; Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (14):
- QGE031 240 mg every 2 weeks (q2w) (Experimental): Participants received QGE031 240 mg subcutaneously (s.c.) q2w for 16 weeks.
  Interventions: Drug: QGE031
- QGE031 240 mg q4w (Experimental): Participants received QGE031 240 mg s.c. q4w for 16 weeks.
  Interventions: Drug: QGE031
- QGE031 180 mg q2w (Experimental): Participants received QGE031 180 mg s.c. q2w for 16 weeks.
  Interventions: Drug: QGE031
- QGE031 120 mg q2w (Experimental): Participants received QGE031 120 mg s.c. q2w for 16 weeks.
  Interventions: Drug: QGE031
- QGE031 36 mg q2w (Experimental): Participants received QGE031 36 mg s.c. q2w for 16 weeks.
  Interventions: Drug: QGE031
- QGE031 12 mg q2w (Experimental): Participants received QGE031 12 mg s.c. q2w for 16 weeks.
  Interventions: Drug: QGE031
- Omalizumab (as per locally approved dosing table) (Active Comparator): Participants received omalizumab as per locally approved dosing table s.c. q2w or q4w for 16 weeks.
  Interventions: Drug: Omalizumab
- Placebo to QGE031 240 mg q2w (Placebo Comparator): Participants received matching placebo to QGE031 240 mg s.c. q2w for 16 weeks.
  Interventions: Drug: Placebo
- Placebo to QGE031 240 mg q4w (Placebo Comparator): Participants received placebo to QGE031 240 mg s.c. q2w for 16 weeks.
  Interventions: Drug: Placebo
- Placebo to QGE031 180 mg q2w (Placebo Comparator): Participants received QGE031 180 mg s.c. q2w for 16 weeks.
  Interventions: Drug: Placebo
- Placebo to QGE031 120 mg q2w (Placebo Comparator): Participants received QGE031 120 mg s.c. q2w for 16 weeks.
  Interventions: Drug: Placebo
- Placebo to QGE031 36 mg q2w (Placebo Comparator): Participants received QGE031 36 mg s.c. q2w for 16 weeks.
  Interventions: Drug: Placebo
- Placebo to QGE031 12 mg q2w (Placebo Comparator): Participants received QGE031 12 mg s.c. q2w for 16 weeks.
  Interventions: Drug: Placebo
- Placebo to omalizumab (Placebo Comparator): Participants received placebo to omalizumab s.c. q2w or q4w for 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QGE031 — QGE031 was supplied as 120 mg liquid in vial per 1 mL
  Arms: QGE031 12 mg q2w; QGE031 120 mg q2w; QGE031 180 mg q2w; QGE031 240 mg every 2 weeks (q2w); QGE031 240 mg q4w; QGE031 36 mg q2w
Drug: Omalizumab — Omalizumab was supplied as 150 mg lyophilisate in vial
  Other Names: Xolair
  Arms: Omalizumab (as per locally approved dosing table)
Drug: Placebo — Placebo to QGE031 and Omalizumab was supplied as QGE031 0 mg in vial per 1 mL
  Arms: Placebo to QGE031 12 mg q2w; Placebo to QGE031 120 mg q2w; Placebo to QGE031 180 mg q2w; Placebo to QGE031 240 mg q2w; Placebo to QGE031 240 mg q4w; Placebo to QGE031 36 mg q2w; Placebo to omalizumab

SUMMARY:
This study assessed the effect on asthma control of different dose levels and regimens of QGE031 in asthma patients that are inadequately controlled with inhaled steroid and beta-2 agonist medication. Safety was assessed also. Comparison was to placebo and omalizumab. Information from this study was planned to support the design of future studies.

ELIGIBILITY:
Key Inclusion Criteria:

* A diagnosis of allergic asthma , uncontrolled on current medication.
* History of at least 1 asthma exacerbation during the last 1 year
* Forced Expiratory Volume in one second (FEV1) of ≥ 40% and ≤ 80% of the predicted normal value; reversibility following administration of bronchodilator must also be demonstrated (historical positive reversibility or bronchoprovocation result can be used).

Key Exclusion Criteria:

* Baseline IgE levels or body weight outside the omalizumab dosing table.
* Use of tobacco products within the previous 6 months (Social occasional smokers may be included).
* Recent asthma attack/exacerbation or asthma worsening/ respiratory infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2012-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (128):
- United States (22):
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Hawaiian Gardens, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, San Jose, California
  - Novartis Investigative Site, Vista, California
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Columbia, Maryland
  - Novartis Investigative Site, Waldorf, Maryland
  - Novartis Investigative Site, Novi, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Papillion, Nebraska
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, Mineola, New York
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Lincoln, Rhode Island
  - Novartis Investigative Site, Mt. Pleasant, South Carolina
  - Novartis Investigative Site, Summerville, South Carolina
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Fairfax, Virginia
  - Novartis Investigative Site, Everett, Washington
- Argentina (9):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires F.D.
  - Novartis Investigative Site, Santa Fe, Rosario
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Santa Fe
- Canada (4):
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Saint-Charles-Borromée, Quebec
  - Novartis Investigative Site, Québec
- Czechia (6):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Trutnov, Czech Republic
  - Novartis Investigative Site, Teplice, CZE
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Břeclav
  - Novartis Investigative Site, Tábor
- Finland (3):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- France (4):
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Strasbourg
- Germany (7):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Roth
  - Novartis Investigative Site, Rüdersdorf
- Guatemala (2):
  - Novartis Investigative Site, Guatemala City, GTM
  - Novartis Investigative Site, Guatemala City
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Törökbálint
- India (3):
  - Novartis Investigative Site, Panjim, Goa
  - Novartis Investigative Site, Karamsad, Gujarat
  - Novartis Investigative Site, Dhantoli, Nagpur
- Israel (5):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
- Italy (6):
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Verona, VR
- Mexico (2):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, México, D.F., Mexico City
- Novartis Investigative Site, Panama City, Panama
- Poland (2):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Lodz
- Portugal (4):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Vila Nova de Gaia
- Romania (8):
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Bucharest, District 3
  - Novartis Investigative Site, Constanța, Jud. Constanta
  - Novartis Investigative Site, Bucharest, ROM
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Piteşti
- Russia (10):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Penza
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Yaroslavl
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (8):
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Nitra, Slovak Republic
  - Novartis Investigative Site, Bardejov
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Prievidza
  - Novartis Investigative Site, Ružomberok
  - Novartis Investigative Site, Trenčín
- South Africa (2):
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Durban
- South Korea (6):
  - Novartis Investigative Site, Bucheon-si, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Cheongju-si, North Chungcheong
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Aydin
  - Novartis Investigative Site, Fatih / Istanbul
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Mersin
- United Kingdom (4):
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, East Yorkshire
  - Novartis Investigative Site, Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 471 participants were randomized to one of the 14 treatment groups. Of these, 5 participants did not receive study treatment. Therefore, the full analysis set (FAS) and safety set included 466 participants.
Pre-assignment Details: The treatment arms for QGE031 and placebo were pooled into high dose QGE031 (240 mg q2w, 240 mg q4w, 180 mg q2w and 120 q2w), low dose QGE031 (36 mg q2w and 18 mg 2qw) and Placebo Total (all QGE031 placebo and Omalizumab placebo arms).
Groups:
- QGE031 High Dose: Participants received QGE031 240 mg q2w, 240 mg q4w, 180 mg q2w or 120 mg q2w.
- QGE031 Low Dose: Participants received QGE031 36 mg q2w or 18 mg q2w.
- Omalizumab: Participants received omalizumab as per locally approved dosing table q2w or q4w.
- Placebo Total: Participants received matching placebo to QGE031 or Omalizumab.
Period: Overall Study
Arm/Group | QGE031 High Dose | QGE031 Low Dose | Omalizumab | Placebo Total
Started | 199 | 40 | 135 | 97
FAS | 199 | 40 | 131 | 96
Safety Set | 199 | 40 | 131 | 96
Completed | 188 | 36 | 121 | 89
Not Completed | 11 | 4 | 14 | 8
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Protocol deviation | 0 | 2 | 7 | 2
Not completed — Non-compliance with study treatment | 0 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Adverse Event | 4 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 5 | 0 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were based on the FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | QGE031 High Dose | QGE031 Low Dose | Omalizumab | Placebo Total | Total
Number analyzed (Participants) | 199 | 40 | 135 | 97 | 471
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.6 (13.86) | 46.0 (12.38) | 46.8 (13.35) | 48.6 (12.80) | 47.4 (13.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 20 | 92 | 63 | 288
  Male | 86 | 20 | 43 | 34 | 183

OUTCOME MEASURES:

1. Primary Outcome: Percentage of QGE031 Participants With Clinically Important Improvement of <= -0.5 in the Asthma Control Questionnaire 7 (ACQ-7) Score Compared to Placebo
Description: The ACQ-7 measures asthma symptom control and consisted of 7 items: 5 on symptom assessment, 1 on rescue bronchodilator use and 1 on airway caliber (FEV1 % predicted). All 7 questions of the ACQ were equally weighted. Items 1-6 scored along a 7-point response scale, where 0 = good controlled and 6 = poor controlled. The 7th item on % predicted FEV1 (pre-bronchodilator) was scored by clinic staff on a 7-point scale (0 - > 95%; 1 - 90-95%; 2 - 80-89%; 3 - 70-79%; 4 - 60-69%; 5 - 50-59%; 6 - < 50%). The average score of the 7 questions was calculated as the sum of scores divided by the number of questions that were answered by the participants, as long as there were at least 6 questions answered and the missing items were neither question 1 nor question 7.
Time Frame: Week 16
Population: The full analysis set (FAS) for the QGE031 240 mg q2w, placebo to QGE031 240 mg q2w and Omalizumab groups (n=120,49,131) was considered for the analysis. Only participants who had week 16 values were analyzed. The FAS included randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Groups:
- QGE031 240 mg q2w: Participants received QGE031 240 mg q2w.
- Placebo to QGE031 240 mg q2w: Participants received placebo to QGE031 240 mg q2w
Arm/Group | QGE031 240 mg q2w | Placebo to QGE031 240 mg q2w | Omalizumab
Number analyzed (Participants) | 114 | 49 | 131
Percentage of participants | 63.16 | 70.21 | 69.17
Statistical Analysis 1: Comparison: QGE031 240 mg q2w vs Placebo to QGE031 240 mg q2w; Test type: Superiority or Other; p = 0.576, Regression, Logistic; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.35 to 1.78]
Statistical Analysis 2: Comparison: QGE031 240 mg q2w vs Omalizumab; Test type: Superiority or Other; p = 0.556, Regression, Logistic; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.46 to 1.52]

2. Secondary Outcome: Change From Baseline in ACQ-7 Score
Description: The ACQ-7 measures asthma symptom control and consisted of 7 items: 5 on symptom assessment, 1 on rescue bronchodilator use and 1 on airway caliber (FEV1 % predicted). All 7 questions of the ACQ were equally weighted. Items 1-6 scored along a 7-point response scale, where 0 = good controlled and 6 = poor controlled. The 7th item on % predicted FEV1 (pre-bronchodilator) was scored by clinic staff on a 7-point scale (0 - > 95%; 1 - 90-95%; 2 - 80-89%; 3 - 70-79%; 4 - 60-69%; 5 - 50-59%; 6 - < 50%). The average score of the 7 questions was calculated as the sum of scores divided by the number of questions that were answered by the participants, as long as there were at least 6 questions answered and the missing items were neither question 1 nor question 7. A negative change from baseline indicates improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 16 and 28
Population: The FAS for the QGE031 240 mg q2w, placebo to QGE031 240 mg q2w and Omalizumab groups (n=120,49,131) was considered for the analysis. Participants who had values at both baseline and the post baseline time point were analyzed for that post baseline time point. The FAS included randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | QGE031 240 mg q2w | Placebo to QGE031 240 mg q2w | Omalizumab
Number analyzed (Participants) | 120 | 49 | 131
Score on a scale
  Week 4 (n=115,46,122) | -0.51 (0.709) | -0.48 (0.834) | -0.60 (0.705)
  Week 8 (n=110,46,122) | -0.68 (0.678) | -0.62 (0.735) | -0.78 (0.687)
  Week 12 (n=110,46,118) | -0.78 (0.738) | -0.71 (0.724) | -0.83 (0.737)
  Week 16 (n=114,48,120) | -0.75 (0.817) | -0.79 (0.733) | -0.89 (0.734)
  Week 28 (n112,47,115) | -0.62 (0.810) | -0.63 (0.744) | -0.59 (0.842)

3. Secondary Outcome: Percentage of Participants With a Change From Baseline in ACQ-7 Score Less Than -1.1
Description: as for outcome 1
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | QGE031 240 mg q2w | Placebo to QGE031 240 mg q2w | Omalizumab
Number analyzed (Participants) | 114 | 47 | 120
Percentage of participants | 40.35 | 34.04 | 36.67
Statistical Analysis 1: Comparison: QGE031 240 mg q2w vs Placebo to QGE031 240 mg q2w; Test type: Superiority or Other; p = 0.483, Regression, Logistic; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.61 to 2.86]
Statistical Analysis 2: Comparison: QGE031 240 mg q2w vs Omalizumab; Test type: Superiority or Other; p = 0.261, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.79 to 2.44]

4. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (AQLQ) Score
Description: The AQLQ is a 32-item disease specific questionnaire designed to measure functional impairments that are most important to participants with asthma. The 32 items in the AQLQ were divided into four domain-specific scores and a total score as follows: Activity limitations = Mean of Items 1, 2, 3, 4, 5, 11, 19, 25, 28, 31, 32 (11 items); Symptoms = Mean of Items 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 29, 30 (12 items); Emotional function = Mean of Items 7, 13, 15, 21, 27 (5 items); Environmental stimuli = Mean of Items 9, 17, 23, 26 (4 items); and Overall Score = Mean of Items 1 to 32 (32 items). Each item of the AQLQ was equally weighted and scored along a 7-point scale, where 1 indicates maximal impairment and 7 indicates no impairment. Thus, higher scores indicate better asthma-related quality of life. The mean overall score ranged from 1 to 7. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 16, Week 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | QGE031 240 mg q2w | Placebo to QGE031 240 mg q2w | Omalizumab
Number analyzed (Participants) | 114 | 48 | 122
Score on a scale
  Week 16 (n=114,48,122) | 0.53 (0.878) | 0.66 (0.624) | 0.79 (0.853)
  Week 28 (n=114,47,121) | 0.44 (0.899) | 0.63 (0.826) | 0.48 (0.871)

5. Secondary Outcome: Change From Baseline in Mean Number of Puffs of Morning, Evening and Total Daily Asthma Rescue Medication
Description: Participants recorded their use of rescue medication into an electronic diary (eDiary). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 16
Population: The full analysis set (FAS) for the QGE031 240 mg q2w, placebo to QGE031 240 mg q2w and Omalizumab groups (n=120,49,131) was considered for the analysis. Only participants who had both baseline and week 16 values were analyzed. The FAS included randomized participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Number of puffs
Arm/Group | QGE031 240 mg q2w | Placebo to QGE031 240 mg q2w | Omalizumab
Number analyzed (Participants) | 117 | 48 | 122
Number of puffs
  Morning | -0.28 (0.072) | -0.34 (0.113) | -0.39 (0.073)
  Evening | -0.31 (0.082) | -0.33 (0.126) | -0.33 (0.084)
  Overall | -0.56 (0.145) | -0.64 (0.226) | -0.73 (0.148)
Statistical Analysis 1: Comparison: QGE031 240 mg q2w vs Placebo to QGE031 240 mg q2w; Morning; Test type: Superiority or Other; p = 0.604, Repeated measures mixed model
Statistical Analysis 2: Comparison: QGE031 240 mg q2w vs Omalizumab; Morning; Test type: Superiority or Other; p = 0.260, Repeated measures mixed model
Statistical Analysis 3: Comparison: QGE031 240 mg q2w vs Placebo to QGE031 240 mg q2w; Evening; Test type: Superiority or Other; p = 0.937, Repeated measures mixed model
Statistical Analysis 4: Comparison: QGE031 240 mg q2w vs Omalizumab; Evening; Test type: Superiority or Other; p = 0.880, Repeated measures mixed model
Statistical Analysis 5: Comparison: QGE031 240 mg q2w vs Placebo to QGE031 240 mg q2w; Overall daily; Test type: Superiority or Other; p = 0.762, Repeated measures mixed model
Statistical Analysis 6: Comparison: QGE031 240 mg q2w vs Omalizumab; Overall daily; Test type: Superiority or Other; p = 0.408, Repeated measures mixed model

ADVERSE EVENTS:
Arm/Group | QGE031 High Dose | QGE031 Low Dose | Omalizumab | Placebo Total
Serious Adverse Events (participants affected / at risk) | 9/199 | 3/40 | 1/131 | 5/96
Other Adverse Events (participants affected / at risk) | 91/199 | 17/40 | 43/131 | 35/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QGE031 High Dose (N=199) | QGE031 Low Dose (N=40) | Omalizumab (N=131) | Placebo Total (N=96)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Vaginal laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Laryngeal dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QGE031 High Dose (N=199) | QGE031 Low Dose (N=40) | Omalizumab (N=131) | Placebo Total (N=96)
Injection site reaction (General disorders) | 57 | 5 | 19 | 5
Nasopharyngitis (Infections and infestations) | 16 | 2 | 9 | 9
Viral upper respiratory tract infection (Infections and infestations) | 6 | 2 | 2 | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 44 | 13 | 19 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.